CLINICAL TRIAL: NCT01991925
Title: Implications for Quality of Life and Quality of Care in Patients With Hereditary Haemochromatosis
Status: Withdrawn | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Annick Vanclooster, Nurse, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: UZL-INT-01
Record Dates: First submitted 2013-11-18; First posted 2013-11-25 (Estimated); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Hereditary Haemochromatosis
MeSH Terms: conditions — Hemochromatosis | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- quality of life, quality of care: hereditary haemochromatosis patients
  Interventions: Other: Interviews, questionaires, RAND-modified delphi method round

INTERVENTIONS:
Other: Interviews, questionaires, RAND-modified delphi method round — phase 1: RAND-modified delphi method round with experts in hereditary haemochromatosis phase 2: patient interviews, questionnaires and focus group interviews

SUMMARY:
Patients with hereditary haemochromatosis will be interviewed/questioned about their Quality of life and the delivered quality of care in the hospital.

DETAILED DESCRIPTION:
Patients with hereditary haemochromatosis will be interviewed/questioned about their Quality of life and the delivered quality of care in the hospital during follow-up

ELIGIBILITY:
Inclusion Criteria:

* phase 1: experts in the field of haemochromatosis (hepatologists, hematologists, endocrinologists, general practitioner, nurses, ...)
* phase 2: patients with hereditary haemochromatosis, treatment with phlebotomy since 3 months, Dutch/English speaking

Exclusion Criteria:

* patients with secondary iron overload
* phlebotomy treatment less than 3 months
* language: no Dutch or English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Phase 1: RAND-modified Delphi Method: experts in the field of hereditary haemochromatosis Phase 2: Patients with hereditary haemochromatosis
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-04; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
evaluation of quality of life | after 3 months of treatment
  quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Annick Vanclooster, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams-brabant, Belgium